CLINICAL TRIAL: NCT03615976
Title: Does Arthroscopic Patellar Denervation With High Tibial Osteotomy Improve Anterior Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, muhammad kamel muhammad sayed, dr: muhammad kamel muhammad sayed, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arthroscopy in P.F.O.A
Record Dates: First submitted 2018-04-16; First posted 2018-08-06 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: arthroscopy; Patellofemoral Osteoarthritis
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: It is prospective case series study The aim is to evaluate the effect of arthroscopic denervation of patella In management of ant. Knee after High tibial osteotomy operation in pain reduction, improving knee joint function, quality of life, and deferring arthritic progression
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): group A with patellofemoral pain resistant to medical and physiotherapy assessment by pre operative knee score HIGH TIBIAL osteotomy will be done for all patients with arthroscopic patellar denervation will be done
  Interventions: Procedure: high tibial osteotomy with or without arthroscopic circumpatellar denervation with or without arthroscopic circumpatellar denervation
- GROUP B (Active Comparator): operative group B with patellofemoral pain resistant to medical and physiotherapy assessment by pre operative knee score HIGH TIBIAL osteotomy will be done without arthroscopic patellar denervation
  Interventions: Procedure: high tibial osteotomy with or without arthroscopic circumpatellar denervation with or without arthroscopic circumpatellar denervation

INTERVENTIONS:
Procedure: high tibial osteotomy with or without arthroscopic circumpatellar denervation with or without arthroscopic circumpatellar denervation — Arthroscopy will be done in all cases before osteotomy to assess lat. Comp and grade of patellofemoral O.A Arthroscopic patellar denervation with vaper or diathermy will be done plus open wedge high tibial osteotomy in one group and other group OWHTO only will be done comparing the rustles of two groups to assess the efficacy of this procedure
  followed by an average follow up to 12 months. And follow up( 6th weeks ,3rd month ,6th month , 12th month)
  By clinical examinationan and x-ray and knee scores
  1. Scoring of patellofemoral disorders( Kujala) score
  2. Knee Injury and Osteoarthritis Outcome Score (KOOS)
  Other Names: arthroscopic circumpatellar denervation

SUMMARY:
Arthroscopy will be done in all cases before osteotomy to assess lat. Comp and grade of patellofemoral O.A Arthroscopic patellar denervation with vaper or diathermy will be done plus open wedge high tibial osteotomy in one group and other group OWHTO only will be done comparing the rustles of two groups to assess the efficacy of this procedure

followed by an average follow up to 12 months. And follow up( 6th weeks ,3rd month ,6th month , 12th month)

By clinical examinationan and x-ray and knee scores

1. Scoring of patellofemoral disorders( Kujala) score
2. Knee Injury and Osteoarthritis Outcome Score (KOOS)

DETAILED DESCRIPTION:
* Patellofemoral joint osteoarthritis (P.F.O.A) is a highly prevalent disease and an important source of anterior knee pain and Disability during daily activities (kneeling, squatting, climbing stairs, getting up from low chair.( 3,5)
* Coexisting Patellofemoral osteoarthritis (PFOA) and Tibiofemoral O.A disease is a common radiographic pattern of knee OA observed in older adults with knee pain. In addition, symptomatic disease and reduced function are more likely to be found if radiographic OA changes are present in both the TF and PF compartment also it demonstrates features distinctly different from those observed in Tibiofemoral O.A without presence of Patellofemoral osteoarthritis (PFOA) . More specifically, "Moderate/Severe PFOA" seems to be associated with lower limb impairments of lower knee extension strength and limitations of knee range of motion. (14)

  * (14,6)
* High tibial osteotomy (HTO) with medial opening wedge has gained in popularity over recent years and is used for the treatment of medial compartmental osteoarthritis (OA) but not for anterior knee pain (P.F.O.A). This procedure is appealing because of the high preservation of the knee joint relative to total knee arthroplasty (TKA) or unicompartmental knee arthroplasty (9)
* High tibial osteotomy (HTO) can cause alterations in patellar height (Patella baja) and alignment which can increase contact stress and eventually lead to anterior Knee pain (13,17)
* The findings indicate that anterior knee pain might be due to OA progression in the patellofemoral joint after HTO (11,12)
* Patellofemoral OA and Cartilage injuries in PF joints tended to progress after Open Wedge HTO which proven by second lock arthroscopy. a significant proportion of patients (about 20%) had grade II OA of the patellofemoral joint at final follow-Up 2yrs. (7,8)
* Anterior knee pain also were quite high (28% and 32% in the opening- and closing-wedge groups) after surgery. Although there are several possible causes for anterior knee pain after HTO, such as surgery itself, alteration of patellar alignment, and OA change in the patellofemoral joint ,patients with severe anterior knee pain were found to have grade II patellofemoral OA. (7,8)
* In spite of its high prevalence, treatment of this painful disorder (PFOA) is challenging due to the diversity of causes of the disorder and the lack of knowledge on articular regeneration, little information is available in the literature about the best conservative or surgical treatment options.(3,5)
* Non-operative treatment options for patellofemoral osteoarthritis include patellar bracing, physical therapy intervention, corticosteroid injections, patellar taping, and strengthening of the quadriceps muscle, this is considered a potential short-term fix for many patients. Ultimately, surgical treatment is necessary to provide a long-term solutions. which include Patellofemoral arthroplasty, total knee replacement with patellar resurfacing,(5)
* Arthroscopic circumpatellar denervation, this joint-preserving, minimal invasive technique provides relief of anterior knee pain. Moreover, this technique provide a faster recovery period immediately after surgery and less morbidity (1,18,19) Arthroscopy will be done in all cases before osteotomy to assess lat. Comp and grade of patellofemoral O.A Arthroscopic patellar denervation with vaper or diathermy will be done plus open wedge high tibial osteotomy in one group and other group OWHTO only will be done comparing the rustles of two groups to assess the efficacy of this procedure

followed by an average follow up to 12 months. And follow up( 6th weeks ,3rd month ,6th month , 12th month)

By clinical examinationan and x-ray and knee scores

1. Scoring of patellofemoral disorders( Kujala) score
2. Knee Injury and Osteoarthritis Outcome Score (KOOS)

ELIGIBILITY:
1. Inclusion criteria:

   1. Age 30-60.
   2. Ant. Knee pain PFOA
   3. Mild to moderate tibiofemoral joint O.A
   4. Without involvement of lateral compartment
   5. Range of motion of at least 120° flexion

   7- BMI less than 30
2. Exclusion criteria:

   1. Old Age more than 60 and less than 30.
   2. Advanced cases tibiofemoral O.A which need TKR
   3. Flextion deformity more than 15 degree
   4. Varus degree more than 10 degree
   5. Inflammatory disease, such as rheumatoid arthritis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Effect of Arthroscopic patellar denervation after open wedge high tibial osteotomy regarding anterior knee pain | all study 2 years average follow up up to 12 months for all cases
  The aim is to evaluate the effect of arthroscopic denervation of patella In management of anterior Knee pain after High tibial osteotomy operation
  The effect of denervation was statistically and clinically evaluated using the Knee injury and Osteoarthritis Outcome Score (KOOS) and Kujala (anterior knee pain score) score

OTHER OUTCOMES:
Effect of OWHTO on ant. Knee pain and patellar height | We will compare the score before and after the surgery and check if it is statically significant. Followed by an average follow up to 12 months ( 6th weeks ,3rd month ,6th month , 12th month)
  Effect of OWHTO on patellar height patellar height (alta or baja) may be evaluated by various methods in the lateral x-ray. We used the Insall-Salvati ratio with a normal ratio of 0.8-1.2. This compared the length of the patellar tendon with the patellar height
Effect of post-operative rehab protocol in Assiut hospital university | We will compare the score before and after the surgery and check if it is statically significant.followed by an average follow up to 12 months ( 6th weeks ,3rd month ,6th month , 12th month)
  Effect of post-operative rehab protocol in Assiut hospital university

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Galal Zaki, PROFESSOR, Study Director — ASSIUT HOSPITAL UNIVERSITY
Locations (1):
- Muhammad Kamel, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Zhao G, Liu Y, Yuan B, Shen X, Qu F, Wang J, Qi W, Zhu J, Liu Y. Arthroscopic patelloplasty and circumpatellar denervation for the treatment of patellofemoral osteoarthritis. Chin Med J (Engl). 2015 Jan 5;128(1):79-84. doi: 10.4103/0366-6999.147820. PMID 25563318
- [Background] Ferrari MB, Sanchez G, Chahla J, Moatshe G, LaPrade RF. Arthroscopic Patellar Lateral Facetectomy. Arthrosc Tech. 2017 Mar 20;6(2):e357-e362. doi: 10.1016/j.eats.2016.10.002. eCollection 2017 Apr. PMID 28580253
- [Background] Waryasz GR, McDermott AY. Patellofemoral pain syndrome (PFPS): a systematic review of anatomy and potential risk factors. Dyn Med. 2008 Jun 26;7:9. doi: 10.1186/1476-5918-7-9. PMID 18582383
- [Background] Witvrouw E, Werner S, Mikkelsen C, Van Tiggelen D, Vanden Berghe L, Cerulli G. Clinical classification of patellofemoral pain syndrome: guidelines for non-operative treatment. Knee Surg Sports Traumatol Arthrosc. 2005 Mar;13(2):122-30. doi: 10.1007/s00167-004-0577-6. Epub 2005 Feb 10. PMID 15703965
- [Background] Wetzels T, Bellemans J. Patellofemoral osteoarthritis treated by partial lateral facetectomy: results at long-term follow up. Knee. 2012 Aug;19(4):411-5. doi: 10.1016/j.knee.2011.04.005. Epub 2011 May 18. PMID 21596570